CLINICAL TRIAL: NCT02829151
Title: Comparison of Cilostazol-based Triple Antiplatelet Therapy Versus Dual Antiplatelet Therapy for Outcomes of below-the Knee Endovascular Intervention in Patients With Critical Limb Ischemia (TAP CLI Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-1104
Record Dates: First submitted 2016-06-20; First posted 2016-07-12 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Critical Limb Ischemia
Keywords: Peripheral artery disease; Critical limb ischemia; Angioplasty; Antiplatelet therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease | interventions — Aspirin; Clopidogrel; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple antiplatelet therapy group (Experimental): Patient group with triple antiplatelet therapy using aspirin, clopidogrel, and cilostazol
  Interventions: Drug: Triple antiplatelet therapy (aspirin (100 mg), clopidogrel (75 mg), and cilostazol (200 mg) )
- DAP (Dual antiplatelet therapy) A (Active Comparator): Patient group with dual antiplatelet therapy using aspirin and clopidogrel
  Interventions: Drug: Dual antiplatelet therapy (aspirin (100 mg) and clopidogrel (75 mg)) using aspirin and clopidogrel
- DAP (Dual antiplatelet therapy) B (Active Comparator): Patient group with angioplasty using aspirin and cilostazol
  Interventions: Drug: Dual antiplatelet therapy (aspirin (100 mg) and cilostazol (200 mg)) using aspirin and cilostazol

INTERVENTIONS:
Drug: Triple antiplatelet therapy (aspirin (100 mg), clopidogrel (75 mg), and cilostazol (200 mg) ) — Combination antiplatelet therapy using aspirin (100 mg), clopidogrel (75 mg), and cilostazol (200 mg) after the index angioplasty
  Arms: Triple antiplatelet therapy group
Drug: Dual antiplatelet therapy (aspirin (100 mg) and clopidogrel (75 mg)) using aspirin and clopidogrel — Combination antiplatelet therapy using aspirin (100 mg) and clopidogrel (75 mg) after the index angioplasty
  Arms: DAP (Dual antiplatelet therapy) A
Drug: Dual antiplatelet therapy (aspirin (100 mg) and cilostazol (200 mg)) using aspirin and cilostazol — Combination antiplatelet therapy using aspirin (100 mg) and cilostazol (200 mg) after the index angioplasty
  Arms: DAP (Dual antiplatelet therapy) B

SUMMARY:
* Prospective, randomized, controlled, multi-center study
* A total of 390 subjects with critical limb ischemia will be included according to inclusion and exclusion criteria.
* Patients will be randomized in a 1:1:1 manner into triple antiplatelet therapy (TAP: aspirin, clopidogrel, cilostazol) group, dual antiplatelet therapy (DAP: aspirin, clopidogrel) A group, or DAP (aspirin, cilostazol) B group.
* All patients will be treated with angioplasty for critical limb ischemia.
* Patients will be followed clinically for 1 year after the procedure.
* Ankle-brachial index and Image study follow-up (Duplex US or CT angiography) will be performed at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 19 years old
* Patients with critical limb ischemia (Rutherford 4 & 5)
* Successful below-the knee endovascular intervention.

Exclusion Criteria:

* Major bleeding event within recent 3 months or high risk of major bleeding
* Patients requiring anticoagulation
* Allergic reactions to antiplatelet drugs
* Acute limb ischemia
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy < 1 year due to comorbidity
* Previous amputations in the target limb

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | 12 months
  A composition event of all-cause death, myocardial infarction, stroke, repeat revascularization of the target lesion, and unexpected amputation of the target limb between TAP group and DAP A group (aspirin & clopidogrel)

SECONDARY OUTCOMES:
Major adverse event between TAP group and DAP B group | 12 months
Adverse limb event among the 3 patient groups | 12 months
Bleeding complications among the patient groups | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided